CLINICAL TRIAL: NCT03544060
Title: Volanesorsen (ISIS 304801) Early Access Program for Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: Volanesorsen Early Access Program for Patients With Familial Chylomicronemia Syndrome (FCS)
Status: No longer available | Type: Expanded Access
Sponsor: Akcea Therapeutics (Industry)
Collaborators: CaligorRx, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: ISIS 304801
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Familial Chylomicronemia
Keywords: Familial Chylomicronemia; Familial Lipoprotein Lipase Deficiency; Hyperlipoproteinemias; Familial Hyperlipoproteinemia Type 1; Hyperlipoproteinemia Type 1; Hyperchylomicronemia, Familial; Lipoprotein Lipase Deficiency, Familial; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Lipid Metabolism, Inborn Errors; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn
MeSH Terms: conditions — Hyperlipoproteinemia Type I; Hyperlipoproteinemias; Familial hyperchylomicronemia syndrome; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Lipid Metabolism, Inborn Errors; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn | interventions — ISIS 304801

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Volanesorsen — Volanesorsen administered by subcutaneous (SC) injections in the abdomen, thigh, or upper arm.
  Other Names: Waylivra

SUMMARY:
The purpose of this program is to provide expanded access to volanesorsen for up to 100 Patients with Familial Chylomicronemia Syndrome (FCS).

DETAILED DESCRIPTION:
The Program is intended to provide expanded access to volanesorsen for eligible patients with FCS who have limited or no available treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the APPROACH Open Label trial, must have completed the open label extension trial for volanesorsen for a length of time consistent with the study protocol (≥ 1 year). Patients in the APPROACH open Label trial for less than a year require approval from Akcea to participate in the EAP. Patients who did not participate in the APPROACH open label trial require approval from Akcea for entry into EAP.
* Patients not participating in the APPROACH open label trial must have a diagnosis of FCS as determined by the participating physician, as outlined in the Volanesorsen EAP protocol. Akcea will review each application to determine eligibility.
* Male patients and female patients of childbearing potential must continue to use appropriate contraception with their partners, or refrain from sexual activity

Exclusion Criteria:

* Patients who have any new conditions or worsening of existing conditions which in the opinion of the Physician would make the patient unsuitable for treatment with volanesorsen.
* Volanesorsen naïve patients with baseline platelet values ≤ 140,000/mm3
* Patients not willing to adhere to mandatory blood draws for platelet monitoring
* Patients who in the opinion of Akcea's medical team, are not eligible candidates for volanesorsen therapy.
* Any patient who plans to or becomes pregnant.
* Any patient who was withdrawn from the APPROACH open label study due to a serious adverse event related to volanesorsen therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult